CLINICAL TRIAL: NCT03881462
Title: Deltoid Muscle Contribution to Shoulder Function - An Experimental Approach
Brief Title: Deltoid Muscle Contribution to Shoulder Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Balgrist University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ID 2019-00135
Record Dates: First submitted 2019-02-15; First posted 2019-03-19 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2019-08

CONDITIONS: Nerve Injury; Nerve Palsy
Keywords: muscle function; rotator cuff

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Axillary nerve block (Experimental): Axillary nerve block is performed in standardized manner and muscle force is measured before and after the block.
  Interventions: Procedure: Axillary nerve block for artificial deltoid muscle palsy

INTERVENTIONS:
Procedure: Axillary nerve block for artificial deltoid muscle palsy — Axillary nerve block block (AXNB):
  The ultrasound probe is placed transversally in the infraclavicular region with the arm in 90° abduction. The brachial plexus and its cords are identified l lateral to the brachial artery. The posterior cord is identified by ultrasound and is blocked - or, if the axillary nerve visible too - the axillary nerve is selectively blocked when it leaves the posterior cord and lies on the subscapular muscle accompanied by the posterior circumflex humeral artery. Using an in-plane technique, a short bevel connected to a nerve stimulator with the setting 0.5 mA current intensity, 0.1 ms impulse duration and 2 Hz impulse frequency for dual guidance, will be advanced until its tip is positioned near the nerve without eliciting motor contractions. After careful negative (for blood) aspiration local anesthetic will be applied until the targeted neuronal structure is surrounded by the injected fluid.

SUMMARY:
There is only one study in the literature about the quantitative effect of M. deltoideus on the movement of the shoulder. Here, the author described a 35-80% loss of abduction power after selective blockade of the N. axillaris. Gerber, on the other hand, found a loss of abduction force of 73-86% after blockade of the suprascapular nerve. These results are partly contradictory, which is why the investigators think that further investigation is needed.

For many questions in the field of shoulder orthopedics, this knowledge would provide an important additional basis for therapeutical decision-making. For example, in the treatment of rotator cuff ruptures but also in the implantation of both inverse and anatomical shoulder prostheses. Also, statements about different outcome prognoses could be made more precisely.

Therefore, the investigators would like to perform muscle strength measurements of the deltoid muscle on 12 healthy volunteers on the dominant arm.

Abduction, flexion, external rotation and internal rotation Mm. Infraspinatus, Supraspinatus and Subscapularis are tested respectively.

The investigators plan to carry out the measurements three times before and after an-anaesthesiological nerve block of the axillary nerve thus inactivating the deltoid muscle (performed exclusively by an anesthesiologist specialized in regional anesthesia). The success of the nerve block is confirmed by needle electromyographies (EMG) by a neurologist specialized in electrophysiology. Using EMG neurogenic pathologies within the tested muscles are also ruled out.

In order to exclude relevant rotator cuff pathologies the investigators will perform shoulder radiography in three planes and sonography of the rotator cuff before conducting the experiment described above.

DETAILED DESCRIPTION:
In order to exclude relevant rotator cuff pathologies the investigators will perform plain shoulder radiography in three planes and sonography of the rotator cuff before conducting the experiment described above.

The force of abduction, flexion, external rotation and internal rotation is measured in a clinically standardized manner with a measuring device (IsoForceControl V1.1) and reported in Newton. These measurements are taken before and after the blockage of the axillary nerve, which is described below. Furthermore, before and after the blockade, an EMG of the rotator cuff and deltoid muscle will be performed in order to rule out neurogenic pathology and confirm the success of the nerve block.

Anesthesia procedure:

In the anesthesia induction area, standard monitoring (electrocardiography, blood oxygen saturation, non-invasive arterial pressure measurement) and peripheral venous access are attained and Ringer's solution will be connected to the venous access.

Axillary nerve block block (AXNB):

The AXNB is performed with the participant in the supine position using ultrasound with a 6- to 13-megahertz (MHz) linear probe.

The anesthesiologist, wearing a facemask, cap, and sterile surgical gloves after surgical hand disinfection performs skin disinfection with a two-layer application of an alcoholic povidone-iodine solution. Three minutes later, the area of the puncture point will be surrounded with sterile drapes and the ultrasound probe will be covered with a sterile cover to allow sterile skin contact.

The ultrasound probe is placed transversally in the infraclavicular region with the arm in 90° abduction. The brachial plexus and its cords are identified l lateral to the brachial artery. The posterior cord is identified by ultrasound and is blocked - or, if the axillary nerve visible too - the axillary nerve is selectively blocked when it leaves the posterior cord and lies on the subscapular muscle accompanied by the posterior circumflex humeral artery. Using an in-plane technique, a short bevel needle (UPC 90, Te-mena) connected to a nerve stimulator with the setting 0.5 milliampere (mA) current intensity, 0.1 ms impulse duration and 2 Hz impulse frequency for dual guidance, will be advanced until its tip is positioned near the nerve without eliciting motor contractions. After careful negative (for blood) aspiration local anesthetic will be applied until the targeted neuronal structure is surrounded by the injected fluid.

In the case of insufficient visualization of the nerve structures with this approach, the investigators will use a modified technique: the volunteer is placed in the sitting position, the shoulder in the neutral position but rotated 45° inward and the elbow flexed at 90° while the hand rested on the knees. Using an in-plane caudad-to-cephalad ultrasound probe placement parallel to the longitudinal axis of the shaft of the humerus and approximately 2cm below the postero-lateral part of the acromion on the dorsal side of the arm the investigators will identify the surgical neck and the shaft of the humerus and the cross section of the posterior circumflex humeral artery (PCHA), The axillary nerve is located cranially in close relation to the PCHA. The nerve will be blocked using the same material as mentioned above.All blocks will be performed by an anesthesiologist specialized in regional anesthesia (U.E. and J.A.) under standard monitoring in an anesthesia working area.

Block success is evaluated assessing the degree of sensory block (cold test) over the distribution area of the axillary nerve every 5 min. The degree of motor block will be assessed by active abduction of the arm every 5 min. After a complete axillary nerve block is documented, the electrophysiological and strength tests will be performed.

Peripheral venous line removal and participant ambulation will be performed after complete motor and sensory recovery of the hand and arm.

All participants will be assessed for neurological status of the blocked extremity by the anaesthesiologist prior to discharge and 24h after the regional anaesthesia.

A photo will be taken for documentation of the elevation function. Electromyographic studies will be performed by experienced neurologists certified in clinical neurophysiology (J.R. & M.S.). Needle EMG serves to verify the axillary block in all three portions of the deltoid muscle, to exclude pathology in the rotator cuff muscles and concomitant anaesthesia thereof. Assessment of possible spontaneous activity, recruitment pattern and motor unit potentials will be performed according to standard methods routinely applied in clinical neurophysiology. Patients on therapeutic anticoagulation will be excluded from needle electromyographic assessments.

ELIGIBILITY:
Inclusion:

* American Society of anesthesiologists (ASA) classification I - II, both sexes
* ≥ 18 years old
* < 65 years old
* Written informed consent as documented by signature

Exclusion:

* Severe coagulopathy or intake of anticoagulants
* History of alcohol abuse or the intake of psychotropic drugs
* Pregnancy
* Infection at the injection site or a systemic infection
* Fever of unknown origin
* Motor or sensory abnormalities in the arm
* Any neuromuscular disorders
* significant arthritis or other shoulder joint problems
* Any co-morbidity that interferes with this study (e.g., stroke, pace maker placement, severe ischemia, cardiac disease, etc.)
* inability to provide informed consent or follow simple instructions during experiment
* contraindications for peripheral regional anaesthesia or local an-esthetics used in the study, e.g., known hypersensitivity or allergy to class of drugs or the investigational product

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Muscle strength of the rotator cuff | 6 hours
  Strength of abduction, flexion, external rotation and internal rotation in Mm. infraspinatus, supraspinatus and subscapularis respectively measured in Newton before and after blockade of the N. axillaris.

SECONDARY OUTCOMES:
Geometric shoulder data | 15 minutes
  Analysis of the geometric data of the X-ray images and correlation with the primary outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Balgrist University Hospital, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No